CLINICAL TRIAL: NCT07020975
Title: The Effect of Virtual Reality Application on Anxiety Before and After Embryo Transfer in Infertile Women
Brief Title: Virtual Reality for Anxiety Relief in Infertile Women
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus Aydin University (Other)
Responsible Party: Principal Investigator, NAZLI ÇATAK, Principal Investigator, Cyprus Aydin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025/04.007
Record Dates: First submitted 2025-06-03; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Anxiety; Assisted Reproductive Treatments; Women; VR; Stress; Virtual Goggles; Infertility; Embryo Transfer
Keywords: Anxiety; Assisted Reproductive Treatments; Women; Nurse; VR; Technology; Infertility; Embryo Transfer
MeSH Terms: conditions — Anxiety Disorders; Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group with VR Glasses (Experimental): Forty women will experience a calming ZEN music soundtrack and view natural landscapes through VR glasses both before and after the embryo transfer procedure.
  Interventions: Device: VR Glasses
- Control Group with routine care (No Intervention): Forty women will receive standard routine care before and after the embryo transfer procedure (Explanation of how to use the medication).

INTERVENTIONS:
Device: VR Glasses — VR Glasses is used to help people be in a virtual reality other than their real life. What we use this for; to get away infertile women from her stressfull environment to another virtual reality before their embryo transfer.
  Arms: Intervention Group with VR Glasses

SUMMARY:
This study examines the impact of virtual reality (VR) applications on anxiety levels before and after embryo transfer procedures. The clinical trial will involve 80 participants, aged 18 to 50, who are receiving treatment at a healthcare facility in the Turkish Republic of Northern Cyprus (TRNC). The primary objective is to evaluate the effectiveness of VR as an intervention for reducing anxiety in individuals undergoing assisted reproductive treatments.

DETAILED DESCRIPTION:
This doctoral study aims to evaluate the use of virtual reality (VR) as an innovative, non-invasive intervention for managing anxiety during embryo transfer in assisted reproductive technology (ART). A randomized clinical trial will be conducted with 80 participants, aged 18 to 50, undergoing fertility treatment at a healthcare facility in the Turkish Republic of Northern Cyprus (TRNC).

Participants will be randomly assigned to one of two groups: the intervention group (n=40), which will experience a VR session both before and after the embryo transfer, and the control group (n=40), which will receive standard care without VR. Anxiety levels will be assessed using the State-Trait Anxiety Inventory (STAI) at two time points-pre- and post-embryo transfer.

The primary objective of this study is to determine the effectiveness of VR in reducing procedural anxiety, a factor known to negatively affect patient experience and potentially influence treatment outcomes. The findings are expected to support the integration of patient-centered, technology-enhanced strategies in reproductive healthcare practices.

ELIGIBILITY:
Inclusion Criteria:

* Volunteered to participate in the research,
* 18-50 years old
* No vision and hearing problems,
* Not disoriented in time and place,
* Primary infertile
* Not having communication problem
* Can read & write
* No mental pathological disease

Exclusion Criteria:

* Secondary infertility
* Having experienced bleeding, miscarriage, etc. after embryo transfer,
* Difficulty communicating,
* Problems such as migraine, vertigo, dizziness,
* Patients who wear prescription glasses and have vision problems without glasses
* Refused to participate in the research
* Patients with psychiatric pathology

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since our participants are women undergoing fertility treatments, only female patients who are scheduled for embryo transfer will be included in the study.
Enrollment: 80 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety level of the women who went through embryo transfer. | 1 year
  This study aims to assess the anxiety levels of women who undergo a virtual reality (VR) experience before and after embryo transfer. The participants will be divided into two groups: those who receive relaxing Zen music and view natural landscapes through VR glasses, and those who do not. Anxiety levels will be objectively measured using the State-Trait Anxiety Inventory, both before and after the embryo transfer procedure.

CONTACTS AND LOCATIONS:
Overall Officials: NAZLI CATAK, MSc, Principal Investigator
Locations (1):
- Cyprus Aydin University, Girne Kepuveia, Keryneia, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Palacios A, Hoffman H, Carlin A, Furness TA 3rd, Botella C. Virtual reality in the treatment of spider phobia: a controlled study. Behav Res Ther. 2002 Sep;40(9):983-93. doi: 10.1016/s0005-7967(01)00068-7. PMID 12296495
- [Background] Freeman D, Reeve S, Robinson A, Ehlers A, Clark D, Spanlang B, Slater M. Virtual reality in the assessment, understanding, and treatment of mental health disorders. Psychol Med. 2017 Oct;47(14):2393-2400. doi: 10.1017/S003329171700040X. Epub 2017 Mar 22. PMID 28325167